CLINICAL TRIAL: NCT05455346
Title: Changes in Biceps Femoris Architecture, Hamstrings Eccentric Strength, and Sprint Performance Following Romanian Deadlift vs. Nordic Hamstring Exercise Intervention
Brief Title: Eccentric Training Effects on Hamstrings Structure, Strength, and Sprint Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2022-0763; Protocol Version 2/27/2023 (Other: UW Madison); A176000 (Other: UW Madison)
Record Dates: First submitted 2022-07-07; First posted 2022-07-13 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Exercise Training; Sport; Running; Ultrasound Imaging; Elastography; Healthy
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: Each eligible participant will be block randomized (1:1 allocation) to either the RDL or the NHE intervention group
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Romanian Deadlift (Experimental): The training intervention groups will undergo the same program with the only difference being the interventional hamstring exercise. The program will consist of a 2-week acclimatization period followed by 4-weeks of progressive training. The RDL will be performed with a 6 second eccentric component with the athlete returning to the start position with a maximal concentric hip extension.
  Interventions: Diagnostic Test: Ultrasound imaging; Other: Hamstring Eccentric Strength Testing; Other: Maximal 60 m Sprint; Other: Romanian Deadlift
- Nordic Hamstring Exercise (Active Comparator): The training intervention groups will undergo the same program with the only difference being the interventional hamstring exercise. The program will consist of a 2-week acclimatization period followed by 4-weeks of progressive training. During the acclimatization period, the relative intensity will be lower compared to the 4-week progressive training to ensure each participant performs the exercise with proper technique. During the subsequent progressive training weeks, the participants will perform the NHE without the bands.
  Interventions: Diagnostic Test: Ultrasound imaging; Other: Hamstring Eccentric Strength Testing; Other: Maximal 60 m Sprint; Other: Nordic hamstring exercise

INTERVENTIONS:
Diagnostic Test: Ultrasound imaging — Ultrasound B-mode images will be unilaterally collected from the biceps femoris muscle of the dominant limb for each participant using a commercial ultrasound system and linear array transducer. Standardized image locations will correspond to 33%, 50%, and 67% of the thigh length from the ischial tuberosity.
  Three repeat longitudinal extended-field-of-view images of the entire biceps femoris muscle will be collected for offline analysis for fascicle length, muscle thickness, and pennation angle. Transverse extended-field-of-view images will be captured at the proximal, mid-belly, and distal locations to determine regional anatomical cross-sectional area of the biceps femoris long head muscle.
  To determine changes in tissue stiffness via ultrasound shear wave speed, the same transducer will be placed in the same locations in a longitudinal view. Shear wave maps will be generated by the ultrasound system and shear wave speed measures extracted from the middle of the map.
Other: Hamstring Eccentric Strength Testing — Prior to each test, participants will perform a standardized 5-minute general warm-up followed by a task-specific warm-up including 3 sets of submaximal trials. Load increases (5-20%) will be added for each RDL 3-repetition maximum trial attempt until the participant cannot complete 3 repetitions through the full range of motion using proper technique. A 3-minute rest will be administered between all warm-up and testing sets to allow for full recovery.
  Participants will kneel on a commercial device used to assess maximum eccentric knee flexor strength via uniaxial load cells with their ankles secured into fixed hooks. Participants will slowly lower their torso to the ground with arms crossed across their chest and without bending at the hips or spine. The maximal test will consist of 1 set of 3 maximal repetitions. If participants can control lower themselves to the ground, then they will hold barbell plates (5-10 lb increments) across their chest while performing the NHE.
Other: Maximal 60 m Sprint — Following a standardized warm-up, inertial measurement units (IMUs) will be placed on the sternum, sacrum, and bilaterally on the thighs, legs, and foot. Each participant will perform a total of 3 maximal 60 m sprints from a standing position with 1.5-3 min rest in between each trial to minimize the effects of fatigue.
Other: Romanian Deadlift — The RDL intervention will be performed twice per week for 6 weeks. Participants will hinge at the hips lowering the bar to just below their patella before reversing the movement. The RDL will be performed with a 6 second eccentric component and returning to the start position with a maximal concentric hip extension.
  Other Names: RDL
  Arms: Romanian Deadlift
Other: Nordic hamstring exercise — The NHE will be performed twice per week for 6 weeks. Participants will be instructed to maintain their ankles in a dorsiflexed position, lower themselves as close to the ground as possible at a constant and controlled speed while maintaining a neutral position of the hips and trunk, and to cross their arms in front of their chest.
  Other Names: NHE
  Arms: Nordic Hamstring Exercise

SUMMARY:
The overall goal of this study is to investigate the effects of a 6-week training program between two hamstring exercises-the Romanian deadlift (RDL) and the Nordic hamstring exercise (NHE)-on hamstring strain injury risk factors and sprint performance.

DETAILED DESCRIPTION:
Prior to the intervention, participants will report to the lab on one occasion for baseline assessments. During the baseline visit, a) regional measures of biceps femoris long head fascicle length, pennation angle, muscle thickness, and anatomical cross-sectional area will be determined using ultrasound, b) baseline NHE strength and 3RM for the RDL will be determined, and c) maximal 60 m sprint performance will be measured.

Participants will be randomly assigned to either the RDL or NHE. After randomization, each participant will undergo the 6 week intervention program based upon their group allocation. Exercises will be performed using a 6 second eccentric (i.e., lowering) contraction.

Following the 6 week intervention, participants would return to the lab for post-intervention assessments of regional hamstring morphology and architecture and sprint testing, which would be carried out in the same manner as baseline assessments. Since fascicle length changes are known to return to baseline values within 2 weeks after the cessation of eccentric training, participants will be asked to return to the lab following a 2 week detraining period where final imaging, strength, and sprint performance assessments will be determined.

ELIGIBILITY:
Inclusion Criteria:

* 18-25 years of age
* Have >6 months experience in resistance training

Exclusion Criteria:

* History of hamstring strain injury within the last 12 months
* History of lower extremity surgery
* Current musculoskeletal injury to the lower extremity
* Females who are currently pregnant
* Individuals who indicate they are unwilling to refrain from novel outside training activities
* Individuals who do not complete 75% (9 out of 12) of the training sessions

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Biceps femoris long head fascicle length | Baseline
Biceps femoris long head fascicle length | Post-intervention (6 weeks)
Biceps femoris long head fascicle length | Post 2 week de-training (8 weeks)

SECONDARY OUTCOMES:
Biceps femoris long head pennation angle | Baseline, Post-intervention (6 weeks), Post 2 week de-training (8 weeks)
Biceps femoris long head muscle thickness | Baseline, Post-intervention (6 weeks), Post 2 week de-training (8 weeks)
Biceps femoris long head anatomical cross sectional area | Baseline, Post-intervention (6 weeks), Post 2 week de-training (8 weeks)
Romanian deadlift (RDL) 3-repetition maximal strength | Baseline, Post-intervention (6 weeks), Post 2 week de-training (8 weeks)
  Maximum weight lifted for 3 repetitions during the RDL
Nordic hamstring exercise (NHE) maximal strength | Baseline, Post-intervention (6 weeks), Post 2 week de-training (8 weeks)
  Maximal eccentric force measured by Nordbord device during NHE
Maximal 60 m sprint times | Baseline, Post-intervention (6 weeks), Post 2 week de-training (8 weeks)
  Fastest 60 m sprint times with interval split times

OTHER OUTCOMES:
Biceps femoris long head regional shear wave speed | Baseline, Post-intervention (6 weeks), Post 2 week de-training (8 weeks)
Inertial measurement unit (IMU)-derived trunk, hip, knee, and ankle kinematics | Baseline, Post-intervention (6 weeks), Post 2 week de-training (8 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Scott K Crawford, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crawford SK, Sandberg C, Vlisides J, Thompson Q, Mosiman SJ, Heiderscheit BC, Hickey JT. Hamstrings Muscle Architecture and Morphology Following 6 wk of an Eccentrically Biased Romanian Deadlift or Nordic Hamstring Exercise Intervention. Med Sci Sports Exerc. 2025 Aug 1;57(8):1799-1809. doi: 10.1249/MSS.0000000000003701. Epub 2025 May 14. PMID 40085810
- [Derived] Crawford SK, Hickey J, Vlisides J, Chambers JS, Mosiman SJ, Heiderscheit BC. The effects of hip- vs. knee-dominant hamstring exercise on biceps femoris morphology, strength, and sprint performance: a randomized intervention trial protocol. BMC Sports Sci Med Rehabil. 2023 Jun 26;15(1):72. doi: 10.1186/s13102-023-00680-w. PMID 37365624